CLINICAL TRIAL: NCT02409446
Title: Metabolic, Vascular and Cognitive Effects of Treatment With Anthocyanins in Older Adults at Risk for Adverse Outcomes - a Pilot Study
Brief Title: Metabolic, Vascular and Cognitive Effects of Treatment With Anthocyanins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Antho 030
Record Dates: First submitted 2015-03-17; First posted 2015-04-06 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2017-12

CONDITIONS: Coronary Disease; Inflammation; Cognitive Impairment
MeSH Terms: conditions — Coronary Disease; Inflammation; Cognitive Dysfunction | interventions — Anthocyanins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anthocyanin (Experimental): 34 patients will receive anthocyanin. We will analyze their blood samples both prior and after taking anthocyanin.
  Interventions: Dietary Supplement: Anthocyanin
- Controls (No Intervention): Healthy Controls, 20 persons. Will be giving blood samples at study start and study end.

INTERVENTIONS:
Dietary Supplement: Anthocyanin — Open pilot study. 35 patients will receive anthocyanin 160 mg x 2 p.o for 16 weeks
  Other Names: Medox
  Arms: Anthocyanin

SUMMARY:
The purpose of this study is to examine weather treatment with anthocyanins will affect lipid profile, markers of inflammation and oxidative stress in addition to antioxidative level in serum to the better in persons with increased risk of dementia.

The purpose of this study is to examine weather treatment with anthocyanins will increase the score of relevant tests of cognitive function.

The investigators will do an open pilot study where patients receive anthocyanin for 16 weeks. 34 patients are expected to be included.

In addition we will include 20 healthy Controls.

DETAILED DESCRIPTION:
Design, method and material:

The investigators will first do an open pilot study where 30 people will receive anthocyanins for 16 weeks.

The investigators aim to recruit persons with increased risk of cognitive reduction: persons over 50 years with stable coronary heart disease (CAD) from the cardiology department Stavanger University Hospital. In addition will persons with mild cognitive impairment or mild dementia be included from the memory outpatient clinic, Stavanger University Hospital.

Blood will be taken by venepuncture by an experienced nurse, centrifuged and handled in according to standardized procedures.

The patients will be tested in relevant tests of cognitive function at inclusion and after 16 weeks. At inclusion the patients will be tested in Mini Mental State Examination (MMSE) and Geriatric depression scale (GDS) to make sure that the patients meet the inclusion criteria. At inclusion and after 16 weeks the patients will be tested in Word List Memory Word List Recall Word List Recognition, Trail Making Test A + B and Stroop Word and Colour test.

From the healthy controls blood will be taken at inclusion and study end.

ELIGIBILITY:
Inclusion Criteria:

* Age above 50 years and coronary suspect chest pain with angiographically CAD without physiologically stenosis
* Mild cognitive impairment (ICD 10) or mild dementia, defined as fulfilling the dementia criteria (ICD 10) but with an MMSE score of 24 or higher.
* Stable medical treatment for the last 3 months.

Exclusion Criteria:

* Moderate to severe dementia (MMSE < 24)
* Clinical significant depression (GDS-15 score of 7 or higher)
* Unstable coronary heart disease
* Heart failure in need of treatment
* Inflammatory illnesses such at rheumatoid arthritis etc.
* Another severe illness with < 5 year expected survival time.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Inflammation as measured by cytokines in blood | 16 weeks
  IL1, IL6, IL10, TNFa
Effect on blood lipids as measured by serum Levels of Cholesterol, triglycerides, cholesterol metabolites | 16 weeks
  Serum Level measurement of Cholesterol, triglycerides, cholesterol metabolites
Effects on oxidative stress as measured by Blood Levels of lipid peroxidation markers, 4-hydroxymenal protein oxydation marker, total protein carbonyl | 16 weeks
  Blood Levels of lipid peroxidation markers, 4-hydroxymenal protein oxydation marker, total protein carbonyl
Effects on antioxidants as measured by Blood levels of vitamin E, vitamin C, vitamin A, total plasma antioxidant capacity, glutathion | 16 weeks
  Blood levels of vitamin E, vitamin C, vitamin A, total plasma antioxidant capacity, glutathion
Number of participants With adverse events | 16 weeks
  Active questioning for adverse events

SECONDARY OUTCOMES:
Effects on memory (CERAD memory test) | 16 weeks
  CERAD memory test, immediate and delayed score
Effects on attention (Trail making A and B) | 16 weeks
  Trail making A and B
Effects on executive functioning (Stroop test) | 16 weeks
  Stroop test
Effects on blood pressure | 16 weeks
  Blood pressure (mm/Hg) in sitting position
Effects on heart rate (ECG) | 16 weeks
  ECG
Effect on Cardiac output (Blood Levels of natriuretic peptides) | 16 weeks
  Blood Levels of natriuretic peptides

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergland AK, Soennesyn H, Dalen I, Rodriguez-Mateos A, Berge RK, Giil LM, Rajendran L, Siow R, Tassotti M, Larsen AI, Aarsland D. Effects of Anthocyanin Supplementation on Serum Lipids, Glucose, Markers of Inflammation and Cognition in Adults With Increased Risk of Dementia - A Pilot Study. Front Genet. 2019 Jun 11;10:536. doi: 10.3389/fgene.2019.00536. eCollection 2019. PMID 31244884